CLINICAL TRIAL: NCT00089349
Title: A Phase II Study of Campath-1H in Children With Acute Lymphoblastic Leukemia in Second or Greater Relapse or Twice Induction Failure
Brief Title: Alemtuzumab With or Without Methotrexate and Mercaptopurine in Treating Young Patients With Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01814; ADVL0222; CDR0000378240; NCI-05-C-0248; COG-ADVL0222; U01CA097452 (NIH); NCT00229606 (obsolete NCT alias)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab; Methotrexate; merphos; Mercaptopurine

ARMS (1):
- Arm I (Experimental): Course 1: Patients receive alemtuzumab IV over 2 hours on days 1-5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission (CR), partial remission (PR), or cytolytic PR at day 29, or patients with CNS disease that achieve a CNS 1 or CNS 2 status, proceed to course 2.
  Courses 2 and 3: Patients receive alemtuzumab IV over 2 hours on days 1, 8, 15, and 22; methotrexate IV continuously over 24 hours on day 1 and then orally once daily on days 8, 15, and 22; and oral mercaptopurine once daily on days 1-28. Patients with a CR or PR at day 29 proceed to course 3. In course 3, patients receive alemtuzumab, methotrexate, and mercaptopurine as in course 2.
  CNS prophylaxis*: Patients receive methotrexate intrathecally on day 1 of courses 2 and 3 on day 1 of courses 2 and 3.
  NOTE: * CNS-negative patients receive methotrexate intrathecally on day 15 of course 1 and day 1 of courses 2 and 3.
  Interventions: Biological: alemtuzumab; Drug: methotrexate; Drug: mercaptopurine

INTERVENTIONS:
Biological: alemtuzumab — Given IV
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: mercaptopurine — Given PO
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP

SUMMARY:
This phase II trial is studying how well giving alemtuzumab with or without methotrexate and mercaptopurine works in treating young patients with relapsed acute lymphoblastic leukemia. Monoclonal antibodies such as alemtuzumab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as methotrexate and mercaptopurine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate to alemtuzumab alone and in combination with methotrexate and mercaptopurine in children with acute lymphoblastic leukemia in second or greater relapse or twice induction failure.

II. Determine the toxicity of these regimens in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of alemtuzumab in these patients. II. Determine the immune response in patients treated with alemtuzumab. III. Determine changes in the number of CD52-positive cells in the blood and marrow of patients treated with alemtuzumab.

IV. Determine the rate and timing of clearance of peripheral circulating lymphoblasts in patients treated with these regimens.

OUTLINE: This is a multicenter study.

Course 1: Patients receive alemtuzumab IV over 2 hours on days 1-5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission (CR), partial remission (PR), or cytolytic PR at day 29, or patients with CNS disease that achieve a CNS 1 or CNS 2 status, proceed to course 2.

Courses 2 and 3: Patients receive alemtuzumab IV over 2 hours on days 1, 8, 15, and 22; methotrexate IV continuously over 24 hours on day 1 and then orally once daily on days 8, 15, and 22; and oral mercaptopurine once daily on days 1-28. Patients with a CR or PR at day 29 proceed to course 3. In course 3, patients receive alemtuzumab, methotrexate, and mercaptopurine as in course 2.

CNS prophylaxis*: Patients receive methotrexate intrathecally on day 1 of courses 2 and 3 on day 1 of courses 2 and 3.

NOTE: * CNS-negative patients receive methotrexate intrathecally on day 15 of course 1 and day 1 of courses 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * Meets 1 of the following criteria:

    * Second or subsequent bone marrow relapse
    * Failed ≥ 2 regimens for remission induction

      * Patients who relapse while receiving standard ALL maintenance chemotherapy do not require a waiting period prior to study entry
* More than 25% blasts in bone marrow aspirate (M3 marrow)

  * CD52 expression on ≥ 25% of malignant cells at relapse
* Philadelphia chromosome-positive patients must have failed prior imatinib mesylate
* Performance status - Karnofsky 50-100% (for patients > 10 years of age)
* Performance status - Lansky 50-100% (for patients ≤ 10 years of age)
* At least 8 weeks
* ALT ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine normal for age
* Pulse oximetry > 94%
* No evidence of dyspnea at rest
* No exercise intolerance
* No serious uncontrolled infection
* No autoimmune hemolytic anemia
* No autoimmune thrombocytopenia
* Not pregnant or nursing

  * No nursing for 3 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* Seizure disorder allowed provided patients are on anticonvulsants and symptoms are well controlled
* CNS toxicity ≤ grade 2
* No other serious uncontrolled medical condition (e.g., diabetes)
* Recovered from prior immunotherapy
* At least 8 weeks since prior biologic agents (e.g., monoclonal antibodies)
* More than 1 week since prior growth factor(s)
* At least 4 months since prior stem cell transplantation

  * No evidence of active acute or chronic graft-versus-host disease post allogeneic stem cell transplantation
* No prior alemtuzumab or its components
* No other concurrent anticancer immunomodulating agents
* Recovered from prior chemotherapy
* One dose of prior intrathecal (IT) methotrexate, cytarabine, and hydrocortisone; IT cytarabine alone; or IT methotrexate alone allowed as part of initial diagnostic spinal tap
* Prior hydroxyurea therapy allowed
* No other concurrent anticancer chemotherapy agents
* Prior steroid therapy allowed
* More than 2 weeks since prior radiotherapy and recovered

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2004-07; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response rate to Campath-1H alone | Day 29, course 1
Response to combined treatment with Campath-1H and chemotherapy | Day 29, course 2
Tolerability of the combination therapy evaluated by dose-limiting toxicity | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Angiolillo, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States